CLINICAL TRIAL: NCT06460363
Title: Transcranial Alternating Current Stimulation on Patients with Delirium and Critical Illness: a Randomized, Controlled, Double Blind, Proof-of-concept Pilot Study
Brief Title: Transcranial Alternating Current Stimulation on Patients with Delirium and Critical Illness (DeliTACS)
Acronym: DeliTACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH507T056
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Delirium
Keywords: Delirium; Tacs; Brain stimulation; Intensive care
MeSH Terms: conditions — Delirium; Spondylocostal Dysostosis 4, Autosomal Dominant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial alternating current stimulation (TACS) (Experimental): Experimental intervention is alternating sinusoidal current at frequency of 40 Hz applied for 60 min through a pair of saline-soaked surface sponge electrodes. One electrode is placed with the center over Pz position according to the 10-20 international EEG coordinates (an area overlying the medial parietal cortex and the precuneus) and the other over the right deltoid muscle.
  Interventions: Device: Transcranial alternating current stimulation (TACS)
- Sham TACS (Sham Comparator): The same electrodes are connected to the patient as in trial intervention. In sham treatment, a few seconds of actual current is provided and then the device automatically turns off. This is to ensure that patients cannot distinguish between real and sham treatments based on possible tingling of skin when starting the electrical current.
  Interventions: Device: Sham TACS

INTERVENTIONS:
Device: Transcranial alternating current stimulation (TACS) — Transcranial alternating sinusoidal current at frequency of 40 Hz applied for 60 min through a pair of saline-soaked surface sponge electrodes.
  Arms: Transcranial alternating current stimulation (TACS)
Device: Sham TACS — Sham treatment with few seconds of actual electrical current and same electrode configuration
  Arms: Sham TACS

SUMMARY:
The goal of this clinical trial is to learn if transcranial alternating current stimulation can shorten the duration of delirium in intensive care setting. The main question it aims to answer:

* Is it possible to shorten the duration of delirium with transcranial alternating current stimulation?

Researchers will compare experimental treatment to sham.

Participants will receive experimental or sham treatment on maximum of two days depending on their delirium status. Duration of delirium is recorded and reported as "days alive and free of delirium".

DETAILED DESCRIPTION:
Delirium is an acute-onset brain dysfunction related to extensive surgery or critical illness that leads to altered mental status and cognitive deficits. Delirium is associated with an increased length of stay in the ICU, cost of care, excessive mortality, and long-term cognitive and functional impairment. Although numerous prophylactic methods have been proposed, currently, no pharmacological or non-pharmacological methods are clinically effective. Patients with delirium have altered electroencephalography (EEG) findings among which most important are general slowing of EEG frequencies and dysconnectivity. Faster EEG frequencies, especially alpha-, beta-, and gamma-bands, are correlated with higher cognitive functions, such as memory and orientation. Transcranial alternating current stimulation (TACS) is a novel, noninvasive brain stimulation technology that cab modulate EEG frequencies by entraining of endogenous brain oscillations in response to exogenous stimuli. TACS has been shown to improve episodic memory, orientation, and cholinergic dysfunction in patients with Alzheimer's disease. TACS also increases alpha and gamma frequencies in EEG, and an increase in these frequencies is associated with the improvement of clinical symptoms. TACS has been shown to target key components of delirium pathophysiology, such as slowing of EEG frequencies and cholinergic dysfunction. Thus, we hypothesized that TACS could shorten the duration of delirium and decrease cognitive decline. We aim to test this hypothesis in a double-blind randomized trial and assess the effect of TACS on duration of delirium, EEG, biomarkers and long-term cognition.

ELIGIBILITY:
Inclusion Criteria:

* Delirium in intensive care and duration of delirium for more than 24 hours. Delirium is defined as 4 or more points on ICDSC and -1 or more points on RASS.

Exclusion Criteria:

* Under 18 years of age, pregnancy, delirium tremens, epilepsy or history of seizures any time before first trial intervention, active psychotic disease, infection of central nervous system, acute intoxication, traumatic brain injury, stroke, intracranial bleeding and implanted electronic devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Days alive and free of delirium or coma | 28 days
  Days alive and free of delirium or coma

SECONDARY OUTCOMES:
Biomarker profile | 4 days
  Concentrations of neurofilament light (nfl), glial fibrillary acid (gfap) and plasma tau (ptau) on days 0, 2 and 4
EEG changes | 2 days
  EEG Spectral power
CERAD | 3 and 12 months
  CERAD test (Consortium to Establish a Registry for Alzheimer's Disease)
TMT test A | 3 and 12 months
  Trail Making Test A
TMT test B | 3 and 12 months
  Trail Making Test B
Short latency inhibition | 3 and 12 months
  Measurement of brain cholinergic function by short latency inhibition with transcranial magnetic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Stepani Bendel, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No